CLINICAL TRIAL: NCT00223561
Title: A Double Blind, Placebo-Controlled Crossover Study to Determine the Effects of Methylphenidate on Driving Ability in Adult Patients With Attention-Deficit Hyperactivity Disorder
Brief Title: Methylphenidate and Driving Ability in Adult Patients With Attention-Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 02/021
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-03-01 (Estimated); Status verified 2006-02

CONDITIONS: ADHD
Keywords: adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: methylphenidate

SUMMARY:
The primary purpose of this study is to determine the effects of methylphenidate versus placebo on driving ability of adult ADHD patients.

DETAILED DESCRIPTION:
This study was set-up to examine the controversial issue whether or not it is safe to drive a car or not when treated with methylphenidate.

On-the-road driving tests during normal traffic are conducted to determine the effects of methylphenidate versus placebo on driving ability of adult ADHD patients.In addition, two laboratory tests are conducted to examine memory functioning and inhibitory control.

ELIGIBILITY:
Inclusion Criteria:

* adult ADHD patient over 21 years old
* valid driver's license for at least 3 years
* treated with methylphenidate
* written informed consent

Exclusion Criteria:

* use of illicit drugs
* use of drugs or having medical conditions known to affect driving ability

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18
Dates: Start 2003-02; Study Completion 2006-02

PRIMARY OUTCOMES:
Driving test:Standard Deviation of Lateral Position (SDLP, cm);i.e. the weaving of the car [single dose effects]

SECONDARY OUTCOMES:
Other Driving test parameters: Standard Deviation of Speed, mean speed, mean lateral position.
Memory test: immediate & delayed word recall, delayed recognition.[single dose effects]
Continuous Performance test: RT, %errors [single dose effects]

CONTACTS AND LOCATIONS:
Overall Officials: Joris Verster, PhD, Principal Investigator — Utrecht Institute for Pharmaceutical Sciences; Edmund Volkerts, PhD, Study Director — Utrecht Institute for Pharmaceutical Sciences
Locations (1):
- Utrecht Institute for Pharmaceutical Sciences, Utrecht, Netherlands

REFERENCES:
- [Derived] Verster JC, Bekker EM, Kooij JJ, Buitelaar JK, Verbaten MN, Volkerts ER, Olivier B. Methylphenidate significantly improves declarative memory functioning of adults with ADHD. Psychopharmacology (Berl). 2010 Oct;212(2):277-81. doi: 10.1007/s00213-010-1952-2. Epub 2010 Jul 20. PMID 20645078